CLINICAL TRIAL: NCT03864536
Title: A Multidomain Approach to Preventing Dementia in African Americans: Cognitive Prescriptions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Pariya L. Fazeli, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Cognitive Prescriptions
Record Dates: First submitted 2019-02-28; First posted 2019-03-06 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Cognitive Change; Health Behavior; Health Literacy
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: A pre-post experimental design will be used, in which 150 AA participants aged 50-65 will complete a baseline assessment of cognitive testing and data-driven assessment of deficiencies across five CogRx domains (physical activity, cognitive activity, diet, sleep, social activity). Participants will be randomized to either: psychoeducation + CogRx, psychoeducation only, or no-contact control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No-contact control (No Intervention): No-contact control
- Psychoeducation control (Active Comparator): Receives general psychoeducation on dementia prevalence, prognosis, and risk factors,
  Interventions: Behavioral: Cognitive Prescriptions
- Psychoeducation + CogRx (Experimental): Receives same general psychoeducation on dementia and will also receive personalized information on their risk factor profile and develop a tailored 3-month intervention plan, which will consist of simple evidence-based strategies to implement at home.
  Interventions: Behavioral: Cognitive Prescriptions

INTERVENTIONS:
Behavioral: Cognitive Prescriptions — Personalized information on their risk factor profile across five CogRx domains (physical activity, cognitive activity, diet, sleep, social activity) and develop a tailored 3-month intervention plan, which will consist of simple evidence-based strategies to implement at home.
  Other Names: CogRx
  Arms: Psychoeducation + CogRx; Psychoeducation control

SUMMARY:
The goal of this R21 study is to explore the feasibility and preliminary efficacy of individualized cognitive prescriptions (CogRxs) in improving engagement in healthy behaviors and other outcomes in middle-aged AAs and to gain feedback on future implementation of the program.

DETAILED DESCRIPTION:
A pre-post experimental design will be used, in which 150 AA participants aged 50-65 will complete a baseline assessment of cognitive testing and data-driven assessment of deficiencies across five CogRx domains (physical activity, cognitive activity, diet, sleep, social activity). Participants will be randomized to either: psychoeducation + CogRx, psychoeducation only, or no contact control. The psychoeducation and CogRx groups will receive general psychoeducation on dementia prevalence, prognosis, and risk factors, while the CogRx group will also receive personalized information on their risk factor profile and develop a tailored 3-month intervention plan, which will consist of simple evidence-based strategies to implement at home. Motivational reminders as well as adherence and self-efficacy questions will be administered via text-messaging over the 3-months. Participants will return for 3-month and 6-month follow-ups. Specific Aim 1 (proximal outcomes) is to determine whether the CogRx condition is superior to psychoeducation alone in improving engagement in healthy lifestyle behaviors. Specific Aim 2 (distal outcomes) is to compare the three conditions on a brief battery of cognitive and psychological measures. The Exploratory Aim is to gather feedback for future implementation of this program, including cultural considerations, barriers and facilitators to engagement, and likelihood of continuing the program.

ELIGIBILITY:
Inclusions:

* Must be African American
* Must be age 50 to 65
* Must have a working cell phone with unlimited texting
* Must be ambulatory

Exclusions:

* No neurological (including dementia diagnosis) or severe psychiatric (e.g., schizophrenia or bipolar disorder) disorders
* No insomnia
* Telephone Interview for Cognitive Status (TICS) score ≤20

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pariya Wheeler, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- the Holly Mears Building/Center for Research on Applied Gerontology, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fazeli PL, Hopkins C, Vance DE, Wadley V, Li P, Turan B, Wang DH, Bowen PG, Clay OJ. Cognitive prescriptions for reducing dementia risk factors among Black/African Americans: feasibility, acceptability, and preliminary efficacy. Ethn Health. 2024 Jan;29(1):1-24. doi: 10.1080/13557858.2023.2231669. Epub 2023 Jul 18. PMID 37463839

RESULTS

PARTICIPANT FLOW:
Groups:
- No-contact Control: No-contact control, has no contact for 3 months
- Psychoeducation Control: Receives general psychoeducation on dementia prevalence, prognosis, and risk factors
Period: Overall Study
Arm/Group | No-contact Control | Psychoeducation Control | Psychoeducation + CogRx
Started | 14 | 12 | 13
Completed | 14 | 12 | 12
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- No-contact Control: No-contact control, no contact for 3 months
- Total: Total of all reporting groups
Arm/Group | No-contact Control | Psychoeducation Control | Psychoeducation + CogRx | Total
Number analyzed (Participants) | 14 | 12 | 13 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (4.6) | 56.0 (6.5) | 55.8 (4.4) | 56.08 (5.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 11 | 32
  Male | 3 | 2 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 12 | 13 | 39
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 13 | 39
TICS-telephone interview for cognitive status [Mean (Standard Deviation); unit: units on a scale] — TICS 11-item measure was used and the total score ranges from 0-41 with higher indicating better cognitive performance. In this study we used the total score, which is a sum across 11 items (each item has a different total possible points).
  units on a scale | 35.2 (3.3) | 33.4 (3.4) | 35.2 (4.0) | 34.67 (3.55)
Marital Status [Count of Participants; unit: Participants]
  In relationship | 3 | 5 | 7 | 15
  Single, Divorced, or Widowed | 11 | 7 | 6 | 24
Employment Status [Count of Participants; unit: Participants]
  Working full or part time | 8 | 9 | 10 | 27
  Not working (unemployed, retired, on disability) | 6 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Leisure Activities Questionnaire Activities Sum
Description: The full measure is a 30-item survey asking about frequency of activities across 4 domains (cognitive, physical, social, and passive), in which higher scores reflect greater engagement in each type of activity (participants rate on Likert scale how often they perform each activity, 0=never/occasionally to 7=daily). The results below reflect a sum of cognitive, physical, and social activities (19 total activities). The total possible sum range is 0 to 133.
Time Frame: change from baseline to 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | No-contact Control | Psychoeducation Control | Psychoeducation + CogRx
Number analyzed (Participants) | 13 | 10 | 12
score on a scale | 1.45 [-5.41 to 8.32] | 4.45 [-3.23 to 12.14] | 11.25 [4.10 to 18.40]
Statistical Analysis 1: Comparison: No-contact Control vs Psychoeducation Control vs Psychoeducation + CogRx; Test type: Superiority; p < 0.05, Mixed Models Analysis — The statistical significance level was set using alpha of 0.05 without multiplicity correction. This pilot study was not powered for all the outcomes so the magnitude and estimates of intervention efficacy was of primary interest

2. Secondary Outcome: Dementia Knowledge
Description: Scores on the Dementia Knowledge Assessment Scale (DKAS-27) which assesses knowledge about risk factors and prognosis of dementia. Scores include percentage correct for the 27 items, with scores ranging from 0-100%. There are 27 items and each item is scored as correct or incorrect. Therefore the scores include a percentage of total items correct, ranging from 0-100 with higher meaning better knowledge.
Time Frame: change from baseline to 3 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | No-contact Control | Psychoeducation Control | Psychoeducation + CogRx
Number analyzed (Participants) | 13 | 10 | 12
score on a scale | 10 [1 to 19] | 27 [16 to 37] | 19 [9 to 28]
Statistical Analysis 1: Comparison: No-contact Control vs Psychoeducation Control vs Psychoeducation + CogRx; Test type: Superiority; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 2 years
Description: This study DSMP stated the PI would serve as the safety officer, given the minimal risk.
Arm/Group | No-contact Control | Psychoeducation Control | Psychoeducation + CogRx
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT03864536/Prot_SAP_000.pdf